CLINICAL TRIAL: NCT05242185
Title: Long Term Sequelae of COVID-19: a Longitudinal Follow-up Study in Dhaka, Bangladesh
Brief Title: Long Term Sequelae of COVID-19: Follow-up Study in Dhaka, Bangladesh
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: PR-20128
Record Dates: First submitted 2022-01-13; First posted 2022-02-16 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19, long term sequelae
MeSH Terms: conditions — COVID-19 | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 survivors: All patients age 18years and more who have SARS-CoV-2 infection confirmed by reverse-transcriptase polymerase-chain-reaction assay (RT-PCR) following their discharge from Dhaka hospital or outpatient clinic or inpatient wards of BSMMU
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — - Baseline data of prognostic importance, including demographic, social information, lifestyle factors, medical history, underlying comorbidities, anthropometric measurements, clinical, laboratory, imaging and treatment records will be collected using a standard case report form. A detailed clinical examination including measurement of vital signs, blood pressure, pulse oximetry, anthropometric measurements, neurological, pulmonary, cardiovascular system examination, mental and fuctional status assessment. routine laboratory assays including complete blood count (CBC), serum alanine transaminase (ALT), serum creatinine, fasting capillary blood glucose using glucometer and urine routine examination, ECG, echocardiography, chest X-ray and pulmonary function test. Additional tests when required such as fasting blood sugar, glycated haemoglobin, MRI/CT scan of brain, Thyroid function tests such as FT4, FT3 and TSH and C peptide etc
  Other Names: Follow- up

SUMMARY:
COVID-19 or coronavirus disease 2019 is an emerging infectious disease. The disease was first identified in China and then spread worldwide; hence, declared as a global pandemic on March 11, 2020 by World Health Organization (WHO). The pandemic is posing formidable challenges to healthcare systems and humanities worldwide resulting in morbidities and mortalities unthought of. Rapidly accumulating clinical evidence on COVID-19 paved the way for an extensive and prompt characterization of the acute phase of the disease. The clinical presentation is generally that of a respiratory infection with a symptom severity ranging from a mild common cold-like illness, to a severe viral pneumonia leading to acute respiratory distress syndrome that is potentially fatal. Characteristic symptoms include fever, cough, and dyspnoea, although some patients may be asymptomatic. Complications of severe disease include, but are not limited to, multi-organ failure, septic shock, and acute respiratory distress syndrome. The COVID-19 infection fatality rate is between 0.5 and 1 percent and the remaining affected patients will mostly recover but need convalescent care. However, discharge should not be considered as the final point of overcoming coronavirus and till date evidence on sequelae of the COVID-19 recovered patients is very limited. COVID-19 is a complex multisystem disease that affects pulmonary function, as well as renal, cardiovascular, and neuropsychiatric health, metabolic derangement; and nutritional status. The extent to which these alterations may persist remains obscure, till date evidence on long term sequelae of the COVID-19 recovered patients is very limited. Some of the aftereffects of it may have a profound impact on 'recovered' patients in the future.

Long-term morbidities were observed in survivors of severe acute respiratory syndrome but it is unidentified whether experience from SARS is applicable to COVID-19. The SARS-CoV-2 infection is severe in older, immune deficient people and who have any pre-existing medical conditions. Hence, it is imperative to comprehend the possible long-term sequelae of the COVID-19 recovered patients, and if they will develop any other harmful illnesses. This study would help us to understand the in-depth prognosis and sequelae of the disease, as well as help to uncover to what extent would COVID-19 recovered patients require post-acute care to recuperate from any further infections or multi-organ damage.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is caused by a novel coronavirus, known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). From December 2019, it has rapidly spread across China and many other countries. COVID-19 pandemic is posing formidable challenges to healthcare systems and humanities worldwide resulting in morbidities and mortalities unthought of.

The first case of COVID-19 was officially detected in Bangladesh on March 8, 2020. As of December 10, 2020, according to the Institute of Epidemiology, Disease Control and Research (IEDCR), there are 485,965confirmed COVID-19 cases in Bangladesh with 6,967 related deaths and the Case Fatality Rate (CFR) is 1.38%. The overall attack rate is 1,639 per 1 million.

Regarding age distribution, 27% of cases were between 31 and 40 years old, 21% in the age group of 21 and 30 years, 19% were between 41 and 50 years, and 15% were in the age group of 51 and 60 years Regarding geographical distribution, 64% of reported confirmed cases were from the Dhaka district, followed by 5.7%in Chattagram district. Case doubling time is 5 days for both the Dhaka and Chattagram district.

COVID-19 is a complex multisystem disease that affects pulmonary function, as well as renal, cardiovascular, and neuropsychiatric health, coagulation derangement as well as nutritional status A significant proportion of patients who survive from COVID-19 may have the possibility to get impairment in their overall health status after their recovery. The extent to which these alterations may persist remains obscure. Some of the aftereffects of it may have a profound impact on 'recovered' patients in the future This study would help us to understand the in-depth prognosis and sequelae of the disease, as well as help to uncover to what extent would COVID-19 recovered patients require post-acute care to recuperate from any further infections or multi-organ damage.

This is a prospective cohort study which will be done in Dhaka hospital of icddr,b and BSMMU. We will include all patients aged ≥ 18 years who have COVID-19, confirmed by reverse-transcriptase polymerase-chain-reaction assay (RT-PCR), following their discharge from Dhaka hospital or outpatient clinic or inpatient wards of BSMMU. Baseline data of prognostic importance, including demographic, social information, lifestyle factors, medical history, underlying comorbidities, anthropometric measurements, clinical, laboratory, imaging and treatment records will be collected using a standard case report form. A detailed clinical examination including measurement of vital signs, blood pressure, pulse oximetry, anthropometric measurements, neurological, pulmonary, cardiovascular system examination will be performed by trained research physicians at enrollment and at each follow-up visit. We will perform routine laboratory assays including complete blood count (CBC), serum alanine transaminase (ALT), serum creatinine, fasting capillary blood glucose using glucometer and urine routine examination. We will also perform ECG, echocardiography, chest X-ray and pulmonary function test. Additional tests will be done as and when required such as RT-PCR test in nasopharyngeal specimen, as well as fasting blood sugar, glycated haemoglobin, MRI/CT scan of brain etc. Thyroid function tests such as FT4, FT3 and TSH and C peptide will be performed at 5 month follow-up time point along with other routine investigations. Participants will be followed up at at 3,5,9,12 ,18 ,24-month time points following discharge from hospital or OPD, and at any time they have a complain.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* Participants categorized as mild, moderate and severe/critical disease according to the classification of WHO and the national guideline on COVID-19 case management published by the DGHS [28], Bangladesh and discharged from the hospital or outpatient clinic
* Participants residing within Dhaka city corporation area
* Willing to participate in this study

Exclusion criteria:

* Participants will be excluded if they have a history mental illness before COVID-19
* Participants with RT-PCR-confirmed SARS-CoV-2 infections but without any relevant clinical symptoms in the preceding fourteen days will be excluded.
* Participants residing outside the Dhaka city corporation area and not willing to participate in the study

Inclusion criteria for comparison group:

Same as exposed group except that they are not exposed to SARS-CoV-2 infection as evident by negative RT-PCR test. Other criteria for comparison group are given below.

* Participants will be included if the RT-PCR test is negative during enrollment
* Age ≥ 18 years
* Participants residing within Dhaka city corporation area
* Willing to participate in this study

Exclusion criteria for comparison group:

• Participants with any known co morbidities including obesity will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include all patients who have SARS-CoV-2 infection confirmed by reverse-transcriptase polymerase-chain-reaction assay (RT-PCR) following their discharge from Dhaka hospital or outpatient clinic or inpatient wards of BSMMU
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-04-04 (Estimated); Study Completion 2022-04-04 (Estimated)

PRIMARY OUTCOMES:
The primary end point will be the prevalence and incidence of long term sequelae of COVID-19 | 24 months
  1. Incidence and prevalence of long-term sequelae
  2. Persistence or development of symptoms at different time-points of follow-up in mild, moderate or severe disease symptoms like
     * dyspnea,
     * fatigue,
     * cough,
     * fever,
     * thoracic pain,
     * nausea,
     * diarrhea,
     * headache

SECONDARY OUTCOMES:
Prevalence and incidence of long term (after 6 weeks) sequelae among OPD and hospitalized group COVID-19 | 24months
  1. Incidence of long term (after 6 weeks) sequelae among survivors of COVID-19
  2. Incidence of abnormal mental health evident by having PTSD as diagnosed by Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) or having a MMSE score of ≤24 (out of 30) or neurological sequelae
  3. Abnormal pulmonary function: Presence of dyspnea as evident by ≥1 score in modified Medical Research Council (mMRC) scale or reduced six-minute walk distance (<580 m men and <500 m for women) or abnormal pulmonary function test.
  4. Cardiovascular sequelae: echocardiographic evidence of pulmonary hypertension and left ventricular dysfunction
  5. New onset diabetes or worsening glycemic control
  6. Incidence of undernutrition, overweight or obesity
  7. Association between demographic, social, lifestyle factors, medical history, underlying comorbidities and persistence of COVID-19 related symptoms and sequelae

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Bangladesh